CLINICAL TRIAL: NCT04736563
Title: Evaluation of the Antalgic Effect of Puressentiel Joints and Muscles - Gel with14 Essential Oils on Joint Pain of the Knee
Brief Title: Evaluation of the Antalgic Effect of Puressentiel Joints and Muscles - Gel on Joint Pain of the Knee
Acronym: EVAPURGEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marco Pacchioni (Industry)
Responsible Party: Sponsor-Investigator, Marco Pacchioni, President Puressentiel laboratory, Puressentiel
Organization: Puressentiel (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Puressentiel laboratory
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pain; Joint Pain
Keywords: Pain; Arthritis; Knee
MeSH Terms: conditions — Pain; Arthralgia; Arthritis

STUDY DESIGN:
Intervention Model Description: open single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with painful arthritis of the knee (Experimental): Administration of joints and muscle gel Puressentiel containing of 14 essential oils
  Interventions: Device: Joint and muscle gel Puressentiel

INTERVENTIONS:
Device: Joint and muscle gel Puressentiel — To evaluate the antalgic effect in patients with chronic pain related to osteoarthritis of the knee when applied to the skin of Puressentiel Joints and Muscles - Gel with 14 essential oils.

SUMMARY:
This clinical trial aims to evaluate the antalgic effect of Puressentiel Joints and Muscles - Gel with 14 essential oils for 12 weeks on knee joint pain in 45 patients suffering from chronic pain related to arthritis of the knee. The evaluation of the puressentiel antalgic effect Joints and Muscles - Gel with 14 essential oils will be done by an algo-functional score of WOMAC based on items of pain, joint stiffness and locomotor function (main criterion), a visual analog scale EVA (graduated from 1 to 10) of the pain by self-assessment of the patient during the consultation and the number of daily analgesics and anti-inflammatory drugs (secondary criteria).

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the antalgic effect of Puressentiel Joints and Muscles - Gel with 14 essential oils for 12 weeks on knee joint pain in 45 patients suffering from chronic pain related to arthritis of the knee. The patients included in the study will be consultants from the Department of Physical Medicine, Rehabilitation and Sports Trauma at Foch Hospital in Suresnes and will have to present chronic pain related to arthritis of the knee either with or without antalgic and anti-inflammatory treatment. The evaluation of the puressentiel antalgic effect Joints and Muscles - Gel with 14 essential oils will be evaluated by an algo-functional score of WOMAC based on items of pain, joint stiffness and locomotor function (main criterion), a visual analog scale EVA (graduated from 1 to 10) of the pain by self-assessment of the patient during each visit and the number of daily antalgic and anti-inflammatory drugs (secondary criteria).

ELIGIBILITY:
Inclusion Criteria:

* Subject smust be able to understand the terms of the written informed consent and must agree to date and sign it before any study procedure is carried out,
* Patient having signed the informed consent
* Aged 45 to 90
* With chronic osteoarthritis of the knee
* Patient with or without analgesic and anti-inflammatory treatment

Exclusion Criteria:

* Patient at the stage of surgical osteoarthritis (grade 4 plus limitation of amplitude)
* Patient with a limited walking perimeter (<100m) for any reason whatsoever
* Patient allergic to one of the components of the study product
* Patient not benefiting from social security
* Patient cannot be followed for the duration of the study
* Participation in another clinical trial within 30 days before V0
* Subjects who cannot understand or perform study procedures.
* Pregnant or breastfeeding women
* People with a history of convulsive or epileptic disorders
* People allergic to salicylates.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Womac score is the primary outcome | 30 days
  Scoring pain and locomotion with a maximum score (worse of 96). A change of 16 points is considered as a significant clinical improvement
Pain visual analog analog scale is the secondary outcome | 30 days
  Scoring pain from 1 to 100 (worse)

SECONDARY OUTCOMES:
Pain visual analog scale | Evaluation at inclusion and after 30 days
  Pain visual analog scale scored from 0 to 100(worse). A change of 10 points is considered as clinically significant

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Simon, Pharm Dr, Study Director — Puressentiel
Locations (1):
- Hopital Foch, Suresnes, France